CLINICAL TRIAL: NCT00574418
Title: Phase 1 Study to Evaluate the Efficacy of Using Energy Specific Far Infrared Radiation Treatment for Uterine Fibroids
Brief Title: Far Infrared Radiation Treatment for Uterine Fibroids
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder & President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-UF-CTP1
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Leiomyoma
Keywords: Fibroid Tumor; Fibroid Uterus; Fibroids, Uterine; Fibromyoma; Uterine Neoplasms
MeSH Terms: conditions — Leiomyoma; Uterine Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Radiation: Far Infrared Radiation (5μm to 20μm wavelength)

INTERVENTIONS:
Radiation: Far Infrared Radiation (5μm to 20μm wavelength) — Far Infrared Radiation (5μm to 20μm wavelength) for 30 to 40 minutes during each session.
  Other Names: Far infrared radiation

SUMMARY:
A preliminary study to determine the efficacy of using energy specific far infrared (FIR) radiation for the treatment of uterine fibroids.

DETAILED DESCRIPTION:
Uterine fibroids are the most common neoplasms of the female pelvis. These benign tumors are generally oval in shape and often highly vascular. On MR imaging exams, uterine fibroids are easily identifiable. They occur in 20-25% of women of reproductive age and can cause a variety of problems generally described as either bleeding or mass effects from the fibroid.

We are postulating that energy specific electromagnetic radiation of the uterus will shrink the benign tumors.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 or older with symptomatic fibroids

Exclusion Criteria:

* Women who are pregnant, as confirmed by serum test at time of screening, or urine pregnancy test on the day of treatment
* Metallic implants that are incompatible with MRI or ultrasound
* Known intolerance to the MRI contrast agent (e.g. Gadolinium)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-01; Primary Completion 2008-03 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
The primary end point is to determine the therapeutic effects of far infrared radiation on uterine fibroids | 2 years and 9 months

SECONDARY OUTCOMES:
The secondary end point of the study is to evaluate the therapeutic effects of far infrared radiation on other related uterine conditions, for example, bleeding. | Two years and nine months

CONTACTS AND LOCATIONS:
Overall Officials: Ken B Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.; Kwasi Donyina, Ph.D., Study Director — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada